CLINICAL TRIAL: NCT04749914
Title: An Open-Label, 2-Part Study to Investigate the Effect of Lasmiditan on the Pharmacokinetics of Dabigatran and Rosuvastatin in Healthy Volunteers
Brief Title: A Study of Lasmiditan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17573; H8H-MC-LAIO (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Drug Interaction Study
MeSH Terms: interventions — lasmiditan; Dabigatran; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 Milligram (mg) Dabigatran Etexilate + 200mg Lasmiditan - Part 1 (Experimental): Participants received 150 mg dabigatran etexilate on Day 1 followed by 200 mg lasmiditan once daily (QD) on Days 8 and 9, and 150 mg of dabigatran etexilate along with 200 mg lasmiditan on Day 10. All treatments were administered orally
  Interventions: Drug: Lasmiditan; Drug: Dabigatran Etexilate
- 10 mg Rosuvastatin + 200 mg Lasmiditan - Part 2 (Experimental): Participants received 10 mg rosuvastatin on Day 1 followed by 200 mg lasmiditan QD on Days 8 and 9, and 10 mg of rosuvastatin along with 200 mg lasmiditan on Day 10. All treatments were administered orally.
  Interventions: Drug: Lasmiditan; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144
Drug: Dabigatran Etexilate — Administered orally.
  Arms: 150 Milligram (mg) Dabigatran Etexilate + 200mg Lasmiditan - Part 1
Drug: Rosuvastatin — Administered orally.
  Arms: 10 mg Rosuvastatin + 200 mg Lasmiditan - Part 2

SUMMARY:
The main purpose of the study is to investigate the blood concentrations of dabigatran etexilate and rosuvastatin when taken alone compared to when taken together with lasmiditan in healthy participants. The safety and tolerability of dabigatran etexilate or rosuvastatin in combination with lasmiditan will also be evaluated in healthy participants. The study has two parts. Each part will last up to 17 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy
* Body mass index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* have known allergies to lasmiditan, dabigatran, rosuvastatin-related compounds or any components of the formulation of lasmiditan, dabigatran, rosuvastatin, or a history of significant atopy
* have an abnormal blood pressure and/or pulse rate as determined by the investigator
* have clinically significant abnormalities on electrocardiogram (ECG) as determined by investigator
* have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study interventions; or of interfering with the interpretation of data. Appendectomy, splenectomy, and cholecystectomy are considered as acceptable
* have any medical conditions, medical history, or are taking any medications that are contraindicated in the dabigatran etexilate or rosuvastatin label
* are intending to use over-the-counter or prescription medication, including dietary supplements, traditional medicines, and herbal supplements, within 14 days prior to dosing and until study discharge (apart from occasional acetaminophen, hormonal contraception, or hormone replacement therapy)
* currently use or show evidence of substance abuse (including alcohol abuse) or dependence within the past 6 months based on history at screening
* Part 1 Only: have known bleeding disorder including prior personal or familial history of abnormal bleeding, hereditary or acquired coagulation or platelet disorder or abnormal coagulation test (prothrombin time/international normalized ratio [INR] or partial thromboplastin time/activated partial thromboplastin time greater than upper limit of normal [ULN]) result at screening
* Part 2 only: have c.34AA, c.421AA, or c.34GA/421CA genotypes of ABCG2 as determined through genotyping

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of two parts - Part 1 and Part 2, each consisting of two periods. Part 1 studied dabigatran P-glycoprotein (P-gp) drug-drug interaction with lasmiditan. Part 2 studied rosuvastatin breast cancer resistance protein (BCRP) drug-drug interaction with lasmiditan.
Groups:
- 150 Milligram (mg) Dabigatran Etexilate-Part 1 Period 1: Participants received a single oral dose 150 mg dabigatran etexilate on Day 1.
- 150 mg Dabigatran Etexilate + 200 mg Lasmiditan-Part 1 Period 2: After Period 1, participants received 200 mg lasmiditan once daily (QD) on Days 8 and 9, and 150 mg of dabigatran etexilate along with 200 mg lasmiditan on Day 10.
- 10 mg Rosuvastatin-Part 2 Period 1: Participants received a single oral dose of 10 mg rosuvastatin on Day 1.
- 10 mg Rosuvastatin + 200 mg Lasmiditan-Part 2 Period 2: After Period 1, participants received 200 mg lasmiditan QD on Days 8 and 9, and then received 10 mg rosuvastatin along with 200 mg lasmiditan on Day 10.
Period: Period 1
Arm/Group | 150 Milligram (mg) Dabigatran Etexilate-Part 1 Period 1 | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan-Part 1 Period 2 | 10 mg Rosuvastatin-Part 2 Period 1 | 10 mg Rosuvastatin + 200 mg Lasmiditan-Part 2 Period 2
Started | 66 | 0 | 31 | 0
Received at Least One Dose of Study Drug | 66 | 0 | 30 | 0
Completed | 64 | 0 | 30 | 0
Not Completed | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Period: Period 2
Arm/Group | 150 Milligram (mg) Dabigatran Etexilate-Part 1 Period 1 | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan-Part 1 Period 2 | 10 mg Rosuvastatin-Part 2 Period 1 | 10 mg Rosuvastatin + 200 mg Lasmiditan-Part 2 Period 2
Started | 0 (Participants who completed Part 1 Period 1 started Part 1 Period 2) | 64 (Participants who completed Part 1 Period 1 started Part 1 Period 2) | 0 (Participants who completed Part 2 Period 1 started Part 2 Period 2) | 30 (Participants who completed Part 2 Period 1 started Part 2 Period 2)
Received at Least One Dose of Study Drug | 0 | 64 | 0 | 30
Completed | 0 | 64 | 0 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- 150 mg Dabigatran Etexilate-Part 1 Period 1: Participants received a single oral dose 150 mg dabigatran etexilate on Day 1.
- Total: Total of all reporting groups
Arm/Group | 150 mg Dabigatran Etexilate-Part 1 Period 1 | 10 mg Rosuvastatin-Part 2 Period 1 | Total
Number analyzed (Participants) | 66 | 30 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 30 | 95
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 6 | 31
  Male | 41 | 24 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 29 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 66 | 30 | 96

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Pharmacokinetics (PK): Maximum Concentration (Cmax) of Dabigatran to Assess P-glycoprotein (P-gp) Activity.
Description: PK: Cmax of Dabigatran.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose.
Population: All participants from Part 1 who received at least 1 dose of Dabigatran etexilate and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 150 mg Dabigatran Etexilate (Part 1 Period 1): Participants received a single oral dose of 150 mg dabigatran etexilate on Day 1.
- 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2): Participants received 200 mg lasmiditan once daily (QD) on Days 8 and 9, and 150 mg of dabigatran etexilate along with 200 mg lasmiditan on Day 10. All treatments were administered orally.
Arm/Group | 150 mg Dabigatran Etexilate (Part 1 Period 1) | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2)
Number analyzed (Participants) | 66 | 64
nanograms/milliliter (ng/mL) | 138 (55) | 168 (51)

2. Primary Outcome: Part 2 PK: Cmax of Rosuvastatin to Assess Breast Cancer Resistance Protein (BCRP) Activity.
Description: PK: Cmax of Rosuvastatin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72 hours post-dose.
Population: All participants from Part 2 who received at least 1 dose of Rosuvastatin and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 10 mg Rosuvastatin (Part 2 Period 1): Participants received a single oral dose of 10 mg rosuvastatin on Day 1.
- 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2): Participants received 200 mg lasmiditan QD on Days 8 and 9, and 10 mg of rosuvastatin along with 200 mg lasmiditan on Day 10. All treatments were administered orally.
Arm/Group | 10 mg Rosuvastatin (Part 2 Period 1) | 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2)
Number analyzed (Participants) | 30 | 30
nanograms per milliliter (ng/mL) | 8.23 (56) | 8.85 (48)

3. Primary Outcome: Part 1 PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞] ) of Dabigatran to Assess P-gp Activity.
Description: PK: AUC[0-∞] of Dabigatran
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose.
Population: All participants from Part 1 who received at least 1 dose of Dabigatran etexilate had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Groups:
- 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2): Participants received 200 mg lasmiditan QD on Days 8 and 9, and 150 mg of dabigatran etexilate along with 200 mg lasmiditan on Day 10. All treatments were administered orally.
Arm/Group | 150 mg Dabigatran Etexilate (Part 1 Period 1) | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2)
Number analyzed (Participants) | 66 | 64
nanogram * hour per milliliter (ng*h/mL) | 1240 (53) | 1540 (50)

4. Primary Outcome: Part 2 PK: AUC[0-∞] of Rosuvastatin to Assess BCRP Activity.
Description: PK: AUC[0-∞] of Rosuvastatin
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72 hours post-dose.
Population: All participants from Part 2 who received at least 1 dose of Rosuvastatin and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Arm/Group | 10 mg Rosuvastatin (Part 2 Period 1) | 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2)
Number analyzed (Participants) | 30 | 30
nanogram * hour per milliliter (ng*h/mL) | 58.6 (60) | 67.3 (52)

ADVERSE EVENTS:
Time Frame: Baseline up to follow up visit, an average of 17 days.
Description: All participants who received at least 1 dose of study drug.
Groups:
- 150 Milligram (mg) Dabigatran Etexilate (Part 1 Period 1): Participants received a single oral dose 150 mg dabigatran etexilate on Day 1.
- 200 mg Lasmiditan (Part 1 Period 2): After Part 1 Period 1, participants received oral doses of 200 mg lasmiditan once daily (QD) on Days 8 and 9.
- 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2): Following lasmiditan administration on Days 8 and 9, participants received 150 mg dabigatran etexilate + 200 mg lasmiditan administered orally on Day 10.
- 200 mg Lasmiditan (Part 2 Period 2): After Part 2 Period 1, participants received oral doses of 200 mg lasmiditan QD on Days 8 and 9.
- 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2): Following lasmiditan administration on Days 8 and 9, participants received 10 mg rosuvastatin + 200 mg lasmiditan administered orally on Day 10.
Arm/Group | 150 Milligram (mg) Dabigatran Etexilate (Part 1 Period 1) | 200 mg Lasmiditan (Part 1 Period 2) | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2) | 10 mg Rosuvastatin (Part 2 Period 1) | 200 mg Lasmiditan (Part 2 Period 2) | 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/64 | 0/64 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/64 | 0/64 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 14/66 | 44/64 | 30/64 | 6/30 | 17/30 | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 Milligram (mg) Dabigatran Etexilate (Part 1 Period 1) (N=66) | 200 mg Lasmiditan (Part 1 Period 2) (N=64) | 150 mg Dabigatran Etexilate + 200 mg Lasmiditan (Part 1 Period 2) (N=64) | 10 mg Rosuvastatin (Part 2 Period 1) (N=30) | 200 mg Lasmiditan (Part 2 Period 2) (N=30) | 10 mg Rosuvastatin + 200 mg Lasmiditan (Part 2 Period 2) (N=30)
Catheter site bruise (General disorders) | 8 (12) | 2 (2) | 11 (13) | 1 (1) | 0 (0) | 1 (2)
Catheter site erythema (General disorders) | 6 (6) | 4 (4) | 4 (4) | 1 (2) | 4 (4) | 3 (3)
Catheter site pain (General disorders) | 8 (8) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 7 (8) | 1 (1) | 6 (7) | 3 (3) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 23 (31) | 7 (7) | 0 (0) | 7 (9) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 9 (10) | 2 (2) | 0 (0) | 7 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT04749914/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04749914/SAP_001.pdf